CLINICAL TRIAL: NCT02816151
Title: Children Toxine Botulinum Detrusor Injection in Neurogenic Vesical Hyperactivity Syndrom: Non Inferiority Multicenter Controlled Therapeutic Study Between Two Reported Weight's Doses
Acronym: TBIDE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PN10002
Record Dates: First submitted 2016-06-24; First posted 2016-06-28 (Estimated); Last update posted 2026-01-21 (Actual); Status verified 2016-06

CONDITIONS: Neurogenic Vesical Hyperactivity Syndrom
MeSH Terms: interventions — abobotulinumtoxinA; Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Group 1 (Experimental)
  Interventions: Drug: full dose at 16 UI/kg for Dysport or 6,5 UA/kg for Botox
- Group 2 (Experimental)
  Interventions: Drug: half dose at 8 UI/kg for Dysport or 3,25 UA/kg for Botox

INTERVENTIONS:
Drug: full dose at 16 UI/kg for Dysport or 6,5 UA/kg for Botox — Intradetrusor injection under general anesthesia. Injection done through 25 points of 1cc each.
  Arms: Group 1
Drug: half dose at 8 UI/kg for Dysport or 3,25 UA/kg for Botox — Intradetrusor injection under general anesthesia. Injection done through 25 points of 1cc each.
  Arms: Group 2

SUMMARY:
Detrusor hyperactivity is an urodynamic observation defined by involuntary detrusor contractions during the vesical filling. Within neurological bladders childs, especially related to spinal dysraphisms, this hyperactivity, associated or not with vesical compliance disorders, can involve a urinary incontinence obstructing social integration and possibly vesical pressure rise in the intra- potentially generating the high urinary tract lesions. Anticholinergic drugs possibly associated with a vesical draining constitute the treatment of first intention. In approximately 15 to 20% of the cases, intradetrusor iterative injections of type A Botulinum Toxin are proposed fault of satisfactory results. Largely used according to the European consensus of 2008 without AM, actual studies remain realized on small numbers with low level of proof. Posology remains discussed between pharmaceutical laboratories (derivative of the effective maximum amount per adult kg of weight) and weaker amounts used with clinical results.

DETAILED DESCRIPTION:
The main aim of the study is to so determine dosages with mid--amount of TBA would make it possible to anticipate not-inferiors results with full posology and to determine the benefit ratio/risk improvement. This could lead to an important reduction of the treatment costs. This study also aims to better identy the "non responders" patients in order to refine the indications. Thanks to the participation of a French urologic paediatric surgery centers, the study hope to homogenize practices and to use standardized common criteria of judgement.

Lastly, this study should appreciate if it is possible not to more bring back posology to the weight of the child, but on detrusor surface allowing a more precise estimation of the amounts to be managed.

A complementary study on the quality of life of these children before and after treatment will be carried out thanks to Child Health Questionnaire (CHQ 50). The diagram of the study is a randomized therapeutic test controlled not-inferiority aiming at comparing an amount full versus an half-amount with TBA.

The population of the study will be made up children from 3 to 15 years treated for detrusor hyperactivity, confirmed by an aurodynamic assessment according to the criteria of International the Society Continence, origin neurological, and resistant to the medical care associated with the usual accompanying measures.

ELIGIBILITY:
inclusion criteria

* Old ≥3 years and ≤15 years
* Syndrome of vesical hyperactivity associated with a manometric detrusor hyperactivity
* Neurogenic vesico-sphincter disorders
* Anticholinergic treatment total/partial Failure/ intolerance
* Native Bladder and TB virgin
* Bladder patient or ready to be it, or possibly straight bladder
* 3 months delay if TB injection in another site
* Agreement to stop anticholinergic treatment 1 month before and throughout all protocol

non- inclusion criteria

* Toxin Botulinic use counter-indication (myasthenia, infantil spinal amyotrophy)
* General anaesthesia counter-indication
* Haemostasis disorders
* Children less than 3 years and more than 16 years
* non-neurogenic vesical hyperactivity
* Good tolerance and effectiveness of the anticholinergic treatment
* Bladder increased or already treated by one or more Toxin injections
* Having toxin injection in another site since less than 3 months
* Child wouldn't sondered

Ages: 3 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 29 (Actual)
Dates: Start 2011-02; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Detrusor pression decrease in neurogenic vesical hyperactivity syndrom for child | up to 6 weeks after intradetrusor injection
  maximal vesical capacity and maximal pression at the end of filling mesured during the course of cystomanometry exam. These points were mesured at leak point or bladder point or when pain appear

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Reims, France, Reims, France

REFERENCES:
- [Background] Leon P, Jolly C, Binet A, Fiquet C, Vilette C, Lefebvre F, Bouche-Pillon-Persyn MA, Poli-Merol ML. Botulinum toxin injections in the management of non-neurogenic overactive bladders in children. J Pediatr Surg. 2014 Sep;49(9):1424-8. doi: 10.1016/j.jpedsurg.2014.04.004. Epub 2014 May 14. PMID 25148752